CLINICAL TRIAL: NCT07228013
Title: Effects of Active Plant Engagement in Campus and Home Environments on College Student Mental Health and Academic Performance
Brief Title: Examining Effects of Active Plant Engagement on College Student Well-Being and Performance
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Responsible Party: Principal Investigator, Kaigang Li, Associate Professor, Director, Colorado State University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 7068
Record Dates: First submitted 2025-11-04; First posted 2025-11-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Perceived Stress; State Anxiety; Intrinsic Goal Orientation; Study Habits; Mood; Sleep Quality; Connectedness to Nature; Extrinsic Goal Orientation
MeSH Terms: conditions — Anxiety Disorders; Sleep Initiation and Maintenance Disorders | interventions — Maintenance

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- G1 (Comparison) (No Intervention)
- G2 (Campus Plant Care) (Experimental): Active care for 1-2 plants in shared academic spaces (e.g. classrooms, hallways)
  Interventions: Behavioral: Active Plant Engagement
- G3 (Home Plant Care) (Experimental): Active care for 1-2 plants in personal living spaces (dorm/apartment)
  Interventions: Behavioral: Active Plant Engagement

INTERVENTIONS:
Behavioral: Active Plant Engagement — Weekly watering, pruning, and soil checks of assigned plants
  Other Names: Hands-on Plant Care and Maintenance
  Arms: G2 (Campus Plant Care); G3 (Home Plant Care)

SUMMARY:
The goal of this feasibility study is to determine if active engagement with plants (e.g. care, maintenance) improves mental health and academic performance in college students. The main questions it aims to answer are:

1. Does active engagement with plants result in improvements in academic motivation and study habits?
2. Does active engagement with plants result in reductions in stress and improvements in mood?

Researchers will compare two interventions groups (campus plant engagement group and home plant engagement group) to the comparison group (no plant engagement or passive exposure) to clarify the practical and potential benefits of active plant care for college students.

Participants will:

* Complete four surveys over the course of a 16-week semester
* Water, prune and check the soil of their assigned plants

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in in-person HES courses during the study semester
* Not currently growing/caring for plants
* Willing to comply with assigned intervention
* Able to complete surveys in English
* Available for 16-week duration

Exclusion Criteria:

* Current enrollment in other intervention studies targeting mental health/academic performance
* Severe plant allergies (e.g. to pollen, mold) regardless of the use of non-toxic and non-pollen plants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2025-08-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Perceived Stress from Baseline to Week 16 | Week 2: Baseline/Time 1 Survey Week 7: Time 2 Survey Week 11: Time 3 Survey Week 16: Time 4 Survey
  The Perceived Stress Scale (PSS) is a validated, widely used measure of stress with clinical relevance in student populations. A significant reduction in Perceived Stress Scale scores would demonstrate a therapeutic effect of the intervention. Scores range from 0-40. Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.
Change in Negative Affect from Baseline to Week 16 | Week 2: Baseline/Time 1 Survey Week 7: Time 2 Survey Week 11: Time 3 Survey Week 16: Time 4 Survey
  The Negative Affect subscale of the Positive and Negative Affect Schedule captures symptoms of anxiety and distress, aligning with the study's focus on mental health. It complements the Perceived Stress Scale by measuring emotional states. Scores of the scale range from 10-50 with higher scores representing higher levels of negative affect.

SECONDARY OUTCOMES:
Change in Sleep Quality from Baseline to Week 16 | Week 2: Baseline/Time 1 Survey Week 7: Time 2 Survey Week 11: Time 3 Survey Week 16: Time 4 Survey
  Assess effects on health behaviors and compare outcomes between communal (campus) vs. personal (home) plant-care environments. Using a single-item self-reported scale to measure sleep quality. Scores range from 0-10. Zero represents 0 hours of quality sleep per night per week and 10 represents 10 hours of quality sleep per night per week. Higher scores indicate better quality of sleep.
Change in Perceived Anxiety from Baseline to Week 16 | Week 2: Baseline/Time 1 Survey Week 7: Time 2 Survey Week 11: Time 3 Survey Week 16: Time 4 Survey
  Assess effects on mental health and well-being using the State Trait Anxiety Inventory to assess acute anxiety reduction. Scores range from 20-80. Scores ranging from 20-37 would be considered low anxiety. Scores from 38-44 would be considered moderate anxiety. Scores from 45-80 would be considered high anxiety.
Change in Perceived Mood Disturbance from Baseline to Week 16 | Week 2: Baseline/Time 1 Survey Week 7: Time 2 Survey Week 11: Time 3 Survey Week 16: Time 4 Survey
  Assess effects on mental health and well-being using the Profile of Moods States scale to assess improvements in tension, depression, and vigor. Scores range from -32 to 200 with higher scores representing a greater degree of overall mood disturbance.
Change in Academic Performance from Baseline to Week 16 | Week 2: Baseline/Time 1 Survey Week 7: Time 2 Survey Week 11: Time 3 Survey Week 16: Time 4 Survey
  Test translational academic performance benefits using self-reported adherence to productive behaviors and the Intrinsic Goal Orientation subscale of the Motivated Strategies of Learning Questionnaire. Scores range from 1-7 with higher scores representing stronger intrinsic goal orientation.
Change in Connectedness to Nature from Baseline to Week 16 | Week 2: Baseline/Time 1 Survey Week 7: Time 2 Survey Week 11: Time 3 Survey Week 16: Time 4 Survey
  Assess effects on health behaviors and compare outcomes between communal (campus) vs. personal (home) plant-care environments. Using a single-item self-reported scale to measure connectedness to nature. 1 represents feelings of no connectedness to nature and 7 represents feelings of high connectedness to nature. Higher scores indicate feelings of a close relationship with nature.

CONTACTS AND LOCATIONS:
Locations (1):
- Colorado State University Health and Exercise Science Department, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van den Bogerd N, Coosje Dijkstra S, Koole SL, Seidell JC, de Vries R, Maas J. Nature in the indoor and outdoor study environment and secondary and tertiary education students' well-being, academic outcomes, and possible mediating pathways: A systematic review with recommendations for science and practice. Health Place. 2020 Nov;66:102403. doi: 10.1016/j.healthplace.2020.102403. Epub 2020 Sep 12. PMID 32932004
- [Background] Jacobson NS, Dobson KS, Truax PA, Addis ME, Koerner K, Gollan JK, Gortner E, Prince SE. A component analysis of cognitive-behavioral treatment for depression. J Consult Clin Psychol. 1996 Apr;64(2):295-304. doi: 10.1037//0022-006x.64.2.295. PMID 8871414
- [Background] Deci EL, Ryan RM. Self-determination theory in health care and its relations to motivational interviewing: a few comments. Int J Behav Nutr Phys Act. 2012 Mar 2;9:24. doi: 10.1186/1479-5868-9-24. PMID 22385839
- [Background] Nuss K, Moore K, Marchant T, Courtney JB, Edwards K, Sharp JL, Nelson TL, Li K. The combined effect of motivational interviewing and wearable fitness trackers on motivation and physical activity in inactive adults: A randomized controlled trial. J Sports Sci. 2023 Jan;41(1):45-55. doi: 10.1080/02640414.2023.2195228. Epub 2023 Mar 25. PMID 36966352
- [Background] Ibrahim AK, Kelly SJ, Adams CE, Glazebrook C. A systematic review of studies of depression prevalence in university students. J Psychiatr Res. 2013 Mar;47(3):391-400. doi: 10.1016/j.jpsychires.2012.11.015. Epub 2012 Dec 20. PMID 23260171
- [Background] Beiter R, Nash R, McCrady M, Rhoades D, Linscomb M, Clarahan M, Sammut S. The prevalence and correlates of depression, anxiety, and stress in a sample of college students. J Affect Disord. 2015 Mar 1;173:90-6. doi: 10.1016/j.jad.2014.10.054. Epub 2014 Nov 8. PMID 25462401
- See also: Bluyssen, PM. (2017). Health, comfort and performance of children in classrooms-new directions for research. Indoor and Built Environment, 26(8), 1040-1050. — https://doi-org.ezproxy2.library.colostate.edu/10.1177/1420326X16661866
- See also: Bringslimark, T, Hartig, T, & Patil, GG. (2007). Psychological benefits of indoor plants in workplaces: Putting experimental results into context. HortScience, 42(3), 581-587. — https://journals-ashs-org.ezproxy2.library.colostate.edu/view/journals/hortsci/42/3/article-p581.xml
- See also: Doxey, JS, Waliczek, TM, & Zajicek, JM. (2009). The impact of interior plants in university classrooms on student course performance and on student perceptions of the course and instructor. HortScience, 44(2), 384-391. — https://journals-ashs-org.ezproxy2.library.colostate.edu/view/journals/hortsci/44/2/article-p384.xml
- See also: Kaplan, R, & Kaplan, S. (1989). The experience of nature: A psychological perspective. Cambridge university press. — https://doi-org.ezproxy2.library.colostate.edu/10.1177/030913259201600333
- See also: Park, S-Y, Song, J-S, Kim, H-D, Yamane, K, & Son, K-C. (2008). Effects of interior plantscapes on indoor environments and stress level of high school students. Journal of the Japanese Society for Horticultural Science, 77(4), 447-454. — http://www.jstage.jst.go.jp.ezproxy2.library.colostate.edu/browse/jjshs
- See also: van den Bogerd, N, Dijkstra, SC, Koole, SL, Seidell, JC, & Maas, J. (2021). Greening the room: A quasi-experimental study on the presence of potted plants in study rooms. Journal of Environmental Psychology, 73, 101557. — https://doi-org.ezproxy2.library.colostate.edu/10.1016/j.jenvp.2021.101557
- See also: Wilson, EO. (1986). Biophilia. Harvard university press. — https://books-google-com.ezproxy2.library.colostate.edu/books?hl=en&lr=&id=gNAuEAAAQBAJ&oi=fnd&pg=PP6&dq=Wilson,+EO.+(1986).+Biophilia.&ots=xw_rRohDCL&sig=ogs9qGT0A4HCB4xPtDICYdNnfNo

DOCUMENTS (1):
  • Informed Consent Form (2025-07-30): https://cdn.clinicaltrials.gov/large-docs/13/NCT07228013/ICF_000.pdf